CLINICAL TRIAL: NCT04583189
Title: Evaluation Des Performances du Test Rapide antigénique Covid-19 Ag BSS Chez l'Enfant Symptomatique Dans un Service d'Urgences pédiatriques
Brief Title: Evaluation of the Performance of the Covid-19 Ag BSS Rapid Antigenic Test in Symptomatic Children in a Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPEEDYCOVI
Record Dates: First submitted 2020-10-01; First posted 2020-10-12 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Covid19
Keywords: Performance of test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test rapid antigenic and Test RT-PCR (Other)
  Interventions: Diagnostic Test: Performance of the test antigenic and test RT-PCR

INTERVENTIONS:
Diagnostic Test: Performance of the test antigenic and test RT-PCR — Each patient will have 1 test rapid antigenic Biosynex Covid-19 Ag-BSS with the results in 15-20 minutes and 1 reference test RT-PCR analyzed in microbiology laboratory of the hospital.

SUMMARY:
This study compares the diagnostic performance of a nasopharyngeal swab antigenic test versus the RT-PCR Covid-19 reference test performed with the AllplexTM 2019-nCoV kit (Seegene, South Korea) in symptomatic children presenting at the hospital.

DETAILED DESCRIPTION:
Since March 2020, France, like the rest of the world, has been suffering from the pandemic caused by SARS CoV-2, which has led to a considerable health crisis. Moreover, the scale of this epidemic was unexpected for the scientific community and the public authorities, who in fact had to find diagnostic and management solutions for COVID-19 most often in the short term. The reference diagnosis of COVID-19 is based on the RT-PCR technique, which allows diagnosis in the early stages of infectious manifestations.

However, since the French recommendations allow widely and without prescription the access the screening of individuals in biology laboratories, regardless of age, symptoms and history of COVID-19 contage, the delays in both the completion of these RT-PCR tests and the return of their results have increased and have become incompatible with relevant decision-making by the clinician and control of the epidemic.

Indeed, since the end of August 2020, it takes about ten days to get the result of an outpatient PCR test. With the increase in the circulation of the SARS-CoV2 virus and the number of positive cases in several regions of France, the use of rapid testing for SARS CoV-2 now seems essential.

Another diagnostic method of COVID-19 is the detection of specific SARS CoV-2 antigens in rhino-pharyngeal secretions and also allows early diagnosis. The qualitative detection of specific SARS CoV-2 antigens by immunochromatography, from rhino-pharynges samples, has the advantage of offering a result in about ten minutes. These tests use specific antibodies from SARS CoV-2 to selectively detect the S protein. Initially these tests like the one developed by the Belgian firm Coris Bioconcept were developed to identify positive COVID-19 patients. Thus, they could be used as rapid screening for screening and would be an alternative to RT-PCR. Their sensitivity varies according to manufacturers and especially according to the viral load between 60% and 90% with a specificity of more than 99%. The sensitivity of this test increases in patients with a high viral load, corresponding to a Ct 25.

In this context of active circulation of the virus and with a Positivity rate in RT-PCR of about 5% in children, it was important for us to evaluate the performance of a rapid diagnostic test by antigenic detection to optimize their management

ELIGIBILITY:
Inclusion Criteria:

*Children under 18 years old requiring an RT-PCR Covid-19 defined according to the algorithm in force at CHI Créteil and which follows the recommendations of the GPIP and the SFP only for symptomatic children :

* Symptomatic children more then 6 years old: cough, and/or fever, and/or digestive disorders unless a diagnosis of another infectious disease is made with certainty (ex Scarlet fever, angina with AMS, enterovirus, urinary tract infections, chickenpox)
* Symptomatic children under 6 years old:

In case of hospitalization or symptoms severe enough to warrant further exploration.

Or who has had a proven contact with a COVID case. Or in contact at home with people considered at risk for SARS-CoV2 infection. Or whose symptoms do not improve after 3 days.

--Febrile children under 3 months old

* Express agreement of one of the parents present, the presence of only one of the two parents being recommanded in the current context
* Affiliated with the Social Security plan

Exclusion Criteria:

Refusal of one of the parents or child to participate in the protocol

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-11-25 (Actual)

PRIMARY OUTCOMES:
Comparison of the performance of the Biosynex Covid-19 Ag BSS rapid antigenic test against the RT-PCR Covid-19 reference test with the AllplexTM 2019-nCoV kit (Seegene, South Korea) in children with symptoms consistent with Covid19 infection | Through study completion up to 30 minutes
  Sensitivity of the Biosynex Covid-19 Ag BSS rapid antigenic test compared to the RT-PCR Covid-19 reference test performed with the AllplexTM 2019-nCoV kit in children.

SECONDARY OUTCOMES:
Sensitivity of the Biosynex Covid-19 Ag BSS rapid antigenic test compared to the RT-PCR Covid-19 reference test performed with the AllplexTM 2019-nCoV kit in children. | Through study completion up to 30 minutes
  -Calculating the entire cohort, based on the age of: Sensitivity, Specificity, Positive predictive value, Negative predictive value, Positive and negative likelihood report Biosynex Covid-19 Ag BSS fast, antigenic test compared to RT-PCR Covid-19 reference test conducted in the laboratory with the AllplexTM 2019-nCoV kit
Comparison of the time it takes to report results between the two methods | Through study completion up to 12 hours
  The difference between the time it takes to allow results between the two types of tests, based on the completion of rhino-pharyngeal tests.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre hospitalier intercommunal de Créteil, Créteil
  - Cabinet de ville, Nogent-sur-Marne
  - Cabinet Dr Cohen, Saint-Maur-des-Fossés
  - Cabinet de ville 13 Villa Beauséjour, Vincennes